CLINICAL TRIAL: NCT02034123
Title: A Phase I Open-label, Dose Escalation Study to Investigate The Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK2879552 Given Orally in Subjects With Relapsed/Refractory Small Cell Lung Carcinoma
Brief Title: Investigation of GSK2879552 in Subjects With Relapsed/Refractory Small Cell Lung Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The risk benefit in relapsed refractory SCLC does not favor continuation of the study
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200858; 2013-003451-38 (EudraCT Number)
Record Dates: First submitted 2013-12-05; First posted 2014-01-13 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Small Cell
Keywords: First time in humans; Small cell lung carcinoma; Oncology; GSK2879552; LSD1 inhibitor
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma; Neoplasms | interventions — GSK2879552

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation Cohort (Experimental): The safety and PK/PD data will be reviewed prior to the dose decision, and the dose escalation will be guided by the Neuenschwander -continuous reassessment method (N-CRM).The dose escalation will complete when RP2D is determined. The RP2D will be the MTD or a lower dose that provides adequate PK exposure and biologic activity with superior tolerability.
  Interventions: Drug: GSK2879552
- Dose Expansion Cohort (Experimental): Once the RP2D has been determined, an expansion cohort of up to 30 subjects will be enrolled in order to better characterize the clinical activity and safety profile of the RP2D
  Interventions: Drug: GSK2879552

INTERVENTIONS:
Drug: GSK2879552 — Subjects will receive GSK2879552orally with approximately 200 milliliter (mL) of water.

SUMMARY:
GSK2879552 is a potent, selective, mechanism-based inactivator of Lysine Specific Demethylase 1 (LSD1)/ CoRepressor for Element-1-Silencing Transcription factor (CoREST) activity. This is a phase I, open-label, multi-center, non-randomized, 2-part first time in human (FTIH) study for GSK2879552. Part 1 is a dose escalation phase to determine the recommended phase 2 dose (RP2D) for GSK2879552 based on the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) profiles observed after oral administration of GSK2879552. Any dose level(s) may be expanded up to 12 subjects in order to collect additional data on PK and PD.The safety and PK/PD data will be reviewed prior to the dose decision, and the dose escalation will be guided by the Neuenschwander -continuous reassessment method (N-CRM). Built-in safety constraints are in place to prevent exposing subjects to undue risk of toxicity. Once RP2D is identified, an expansion cohort (Part 2) of up to 30 subjects will be enrolled to further evaluate the clinical activity and tolerability of GSK2879552 in subjects with relapsed/refractory SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent
* Males and females >=18 years of age (at the time consent is obtained).
* Histologically or cytologically confirmed diagnosis of small cell lung carcinoma. Subjects must have measurable disease per RECIST 1.1 (for Part 2 only).
* Recurrent or refractory disease after receiving at least one prior standard/approved platinum-containing chemotherapy regimen, or where standard therapy is refused. Part 2 only: Subjects must have recurrent disease after receiving a maximum of two prior chemotherapy regimens including at least one platinum containing regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 1. (ECOG performance status of 0 or 1).
* Tumor tissue requirements: Availability of archival tissue, or willingness to undergo fresh biopsy at baseline; Enrollment in PK/PD cohort may be limited to subjects with disease amenable to pre- and post-dose biopsies, and willingness to undergo biopsy.
* All prior treatment-related toxicities must be National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 <=Grade 1 at the time of enrollment (except for alopecia)
* Adequate baseline organ function
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception, as defined in protocol, during the study and for 7 days following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described in protocol from the administration of the first dose of study treatment until 3 months after the last dose of study treatment to allow for clearance of any altered sperm.
* Able to swallow and retain orally administered study treatment and does not have any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Concurrent malignancy other than SCLC. History of other malignancy is allowed as long as there is no evidence of active disease or need for treatment.
* Currently receiving anti-cancer therapy. Exceptions: Zoledronic acid and denosumab to treat bone metastasis are allowed.
* Prior treatment with temozolomide, dacarbazine or procarbazine.
* Prior treatment with poly ADP ribose polymerase (PARP) inhibitors (e.g., olaparib, ABT-888).
* Baseline Montreal Cognitive Assessment (MOCA) score of 22 or lower.
* Received major surgery, radiotherapy, or immunotherapy within 4 weeks of GSK2879552 administration. Chemotherapy regimens with delayed toxicity within the last four weeks (six weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity or palliative radiation to a limited area within the last two weeks.
* Administration of an investigational drug within 28 days or 5 half-lives, whichever is shorter preceding the first dose of study treatment(s) in this study.
* French subjects: The French subject has participated in any study using an investigational study treatment(s) during the previous 28 days.
* Subjects with current/a history of bleeding disorder or coagulopathy or who are at particularly high risk for bleeding complications.
* Requiring anticoagulants at therapeutic doses or platelet inhibitor.
* Current use of a prohibited medication or expected to require any of these medications during treatment with the investigational drug
* Evidence of severe or uncontrolled systemic diseases. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator
* Known active Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infections. Subjects with laboratory evidence of HBV clearance may be enrolled
* Leptomeningeal metastases or spinal cord compression due to disease.
* Subjects with previously untreated or uncontrolled brain metastases.
* Cardiac abnormalities
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2879552 or LSD1 inhibitors that contraindicates their participation.
* Lactating female
* Consumption of Seville oranges, grapefruit, grapefruit hybrids, grapefruit juice, pommelos, or exotic citrus fruits, from 1 day prior to the first dose of study treatment(s) until the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (3):
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Nashville, Tennessee
- GSK Investigational Site, Villejuif, France
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20058

REFERENCES:
- [Background] Bauer TM, Besse B, Martinez-Marti A, Trigo JM, Moreno V, Garrido P, Ferron-Brady G, Wu Y, Park J, Collingwood T, Kruger RG, Mohammad HP, Ballas MS, Dhar A, Govindan R. Phase I, Open-Label, Dose-Escalation Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of GSK2879552 in Relapsed/Refractory SCLC. J Thorac Oncol. 2019 Oct;14(10):1828-1838. doi: 10.1016/j.jtho.2019.06.021. Epub 2019 Jun 28. PMID 31260835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was planned as a 2-part, first time in human study in participants with relapsed/refractory small cell lung carcinoma. Part 1 was a dose escalation cohort and Part 2 was an expansion cohort. Participants were planned to receive GSK2879552 at a starting dose of 0.25 milligrams (mg) once daily for 28 days.
Pre-assignment Details: This study was terminated early during Part 1 as the risk benefit in relapsed refractory SCLC did not favor continuation of the study. Data was collected only in Part 1 and no participants were enrolled in Part 2. A total of 29 participants enrolled and received treatment in Part 1. Of which 7 prematurely withdrawn and 22 completed study.
Groups:
- Part 1:GSK2879552 0.25 mg Daily: Participants received GSK2879552 with a starting dose of 0.25 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1:GSK2879552 0.5 mg Daily: Participants received GSK2879552 with a dose of 0.5 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1:GSK2879552 1.0 mg Daily: Participants received GSK2879552 with a dose of 1.0 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1:GSK2879552 1.5 mg Daily: Participants received GSK2879552 with a dose of 1.5 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1: GSK2879552 2.0 mg Daily: Participants received GSK2879552 with a dose of 2.0 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1: GSK2879552 3.0 mg Daily: Participants received GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off: Participants received GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 3 days.
- Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off: Participants received GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 10 days.
- Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off: Participants received GSK2879552 with a dose of 4.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 10 days.
- Part 2:GSK2879552 0.25 mg Daily: Participants were planned to receive GSK2879552 with a starting dose of 0.25 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2:GSK2879552 0.5 mg Daily: Participants were planned to receive GSK2879552 with a dose of 0.5 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2:GSK2879552 1.0 mg Daily: Participants were planned to receive GSK2879552 with a dose of 1 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2:GSK2879552 1.5 mg Daily: Participants were planned to receive GSK2879552 with a dose of 1.5 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2: GSK2879552 2.0 mg Daily: Participants were planned to receive GSK2879552 with a dose of 2.0 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2: GSK2879552 3.0 mg Daily: Participants were planned to receive GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 28 days.
- Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off: Participants were planned to receive GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 3 days.
- Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off: Participants were planned to receive GSK2879552 with a dose of 3.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 10 days.
- Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off: Participants were planned to receive GSK2879552 with a dose of 4.0 mg once daily, administered orally with approximately 200 milliliter of water for 4 days during the treatment period following buffer period of 10 days.
Period: Part1(Median of 7.286 Weeks of Exposure)
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Started | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 5 | 1 | 5 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other-Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part2(Up to 2 Years)
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected only in Part 1 and no participants were enrolled in Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off | Total
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.0 (NA) — NA indicates data was not available due to insufficient number of participants to calculate standard deviation. | 47.0 (NA) — NA indicates data was not available due to insufficient number of participants to calculate standard deviation. | 63.8 (4.09) | 56.7 (8.08) | 62.4 (7.41) | 60.3 (7.51) | 53.5 (13.44) | 58.8 (10.33) | 61.5 (9.19) |  |  |  |  |  |  |  |  |  | 60.6 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 1 |  |  |  |  |  |  |  |  |  | 11
  Male | 0 | 0 | 4 | 3 | 6 | 1 | 1 | 2 | 1 |  |  |  |  |  |  |  |  |  | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  |  |  |  |  |  |  | 1
  White-White/Caucasian/European Heritage | 1 | 1 | 5 | 3 | 7 | 3 | 1 | 5 | 2 |  |  |  |  |  |  |  |  |  | 28

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. The analysis was performed on All Treated Population which included all participants who received at least one dose of study treatment.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants
  Any non-SAE | 1 | 1 | 5 | 2 | 6 | 3 | 2 | 5 | 1
  Any SAE | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 2

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: An event was considered a DLT if it occurs within the first 28 days of treatment, and meets one of the following criteria unless it can be clearly established that the event is unrelated to treatment: recurrent Grade 3 anemia after initial transfusion or Grade 3 anemia lasting > 7 days in participants who are not transfused, Grade 4 neutropenia, Grade 3 neutropenia > 7 days duration, febrile neutropenia as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, Grade 3 thrombocytopenia requiring dose reduction, Grade 4 thrombocytopenia lasting > 3 days or of any duration if associated with clinically significant bleeding, drug related Grade 3 or 4 non-hematologic toxicity, drug related Grade 2 toxicity (at any time during treatment) and treatment delay of 14 days or greater due to unresolved drug-related toxicity.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0

3. Primary Outcome: Part 1: Number of Participants With Dose Reduction or Delays
Description: The number of participants who had any dose reduction or delay have been presented. All dose reductions were due to AEs.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | 1 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants Withdrawn Due to Toxicities
Description: Participants were monitored from start of the study till the development of toxicity. The data for number of participants withdrawn due to toxicities has been presented.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

5. Primary Outcome: Part 1: Number of Participants With Change in Clinical Chemistry Toxicity Grade From Baseline
Description: Blood samples were collected for evaluation of clinical chemistry parameters including potassium, aspartate aminotransferase (AST), total bilirubin, creatinine, alanine aminotransferase (ALT), uric acid, glucose, gamma glutamyl transferase (GGT), albumin, sodium, calcium, alkaline phosphatase, and phosphorus, inorganic. Baseline value was defined as the most recent, non-missing value from a central laboratory prior to or on the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The number of participants with any grade increase in clinical chemistry parameters have been presented. The clinical chemistry parameters for which any grade increase worst-case on-therapy value was reported have been only summarized. NA represents data was not available. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants
  Albumin;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Albumin;n=1,1,5,3,5,3,2,5,2 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 1
  Alkaline Phosphatase;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Alkaline Phosphatase;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 2 | 0
  ALT;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  ALT;n=1,1,5,3,5,3,2,5,2 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 1
  AST;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  AST;n=1,1,5,3,5,3,2,5,2 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 2 | 1
  Total Bilirubin;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Total Bilirubin;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Calcium;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0
  Calcium (hypercalcemia);n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Calcium (hypercalcemia);n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
  Calcium (hypocalcemia);n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Calcium (hypocalcemia);n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Creatinine;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1
  GGT;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  GGT;n=1,1,5,3,5,3,2,5,2 | 1 | 1 | 4 | 1 | 2 | 3 | 1 | 2 | 1
  Glucose;n=1,1,5,3,6,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 2
  Glucose;n=1,1,5,3,6,3,2,5,2 | 1 | 1 | 2 | 1 | 4 | 1 | 1 | 3 | 1
  Glucose (hyperglycemia);n=1,1,5,3,6,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 2
  Glucose (hyperglycemia);n=1,1,5,3,6,3,2,5,2 | 1 | 1 | 2 | 1 | 4 | 1 | 1 | 3 | 1
  Glucose (hypoglycemia);n=1,1,5,3,6,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 2
  Glucose (hypoglycemia);n=1,1,5,3,6,3,2,5,2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium;n=1,1,5,2,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 2 | 5 | 3 | 2 | 5 | 2
  Potassium;n=1,1,5,2,5,3,2,5,2 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0
  Potassium (hyperkalemia);n=1,1,5,2,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 2 | 5 | 3 | 2 | 5 | 2
  Potassium (hyperkalemia);n=1,1,5,2,5,3,2,5,2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Potassium (hypokalemia);n=1,1,5,2,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 2 | 5 | 3 | 2 | 5 | 2
  Potassium (hypokalemia);n=1,1,5,2,5,3,2,5,2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
  Sodium;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Sodium;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 3 | 0 | 2 | 1 | 1 | 1 | 0
  Sodium (hypernatremia);n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Sodium (hypernatremia);n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Sodium (hyponatremia);n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Sodium (hyponatremia);n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 1 | 0
  Phosphorus, inorganic;n=1,1,5,3,5,3,2,5,2: number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 2
  Phosphorus, inorganic;n=1,1,5,3,5,3,2,5,2 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0
  Uric acid;n=0,0,1,0,0,1,0,0,1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Uric acid;n=0,0,1,0,0,1,0,0,1 |  |  | 1 |  |  | 1 |  |  | 1

6. Primary Outcome: Part 1: Number of Participants With Change in Hematology Toxicity Grade From Baseline
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin, lymphocytes, total neutrophils, platelet count and white blood cell (WBC) count. Baseline value was defined as the most recent, non-missing value from a central laboratory prior to or on the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The number of participants with any grade increase in hematology parameters have been presented. The hematology parameters for which any grade increase worst-case on-therapy value was reported have been only summarized.
Time Frame: Baseline and median of 7.286 weeks of drug exposure
Population: All Treated Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 2
Participants
  Hemoglobin | 1 | 0 | 3 | 2 | 4 | 2 | 0 | 3 | 1
  Hemoglobin (Increased) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (Anemia) | 1 | 0 | 3 | 2 | 4 | 2 | 0 | 3 | 1
  Lymphocytes | 0 | 0 | 3 | 2 | 2 | 2 | 1 | 4 | 1
  Lymphocytes (Increased) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (Decreased) | 0 | 0 | 3 | 2 | 2 | 2 | 1 | 4 | 1
  Total Neutrophils | 1 | 0 | 2 | 0 | 2 | 2 | 2 | 1 | 0
  Platelet count | 1 | 0 | 3 | 1 | 5 | 3 | 1 | 4 | 0
  WBC count | 1 | 0 | 2 | 0 | 2 | 3 | 2 | 3 | 0

7. Primary Outcome: Part 1:Number of Participants With Critical Changes in Values of Vital Signs in Response to Drug
Description: Vital sign measurements includes systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature, respiration rate and heart rate. Vital signs were measured after resting for at least 5 minutes in a semi-supine position. The number of participants with critical changes in values of vital signs in response to drug have been presented.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 1: Number of Participants With Abnormal Findings for Electrocardiogram (ECG) Parameters
Description: Single measurements of 12-lead ECGs were obtained in a semi-recumbent or supine position after at least a 5 minutes rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. The number of participants with abnormal - not clinically significant and abnormal - clinically significant "worst-case on-therapy" value have been presented.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 5 | 3 | 2 | 5 | 1
Participants
  Abnormal - not clinically significant | 0 | 1 | 4 | 1 | 4 | 1 | 1 | 5 | 1
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Abnormal Findings Undergoing Physical Examinations
Description: The complete physical examination included assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. A brief physical examination included assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). All abnormal physical examination findings were reported as AEs within the AE specific case report form (CRF) page. Hence, data was not captured separately for this outcome as number of participants with abnormal findings with respect to physical examinations. NA indicates data was not available as all abnormal physical examination findings were reported as AEs.
Time Frame: Median of 7.286 weeks of drug exposure
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs. | NA — NA indicates data was not available as all abnormal physical examination findings were reported as AEs.

10. Primary Outcome: Part 2: Number of Participants Achieving Disease Control Rate at Week 16
Description: Clinical response was planned to be assessed by the investigator using computer tomography or magnetic resonance imaging scans. Clinical response was defined as disease control rate based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at Week 16. Disease control rate was defined as number of participants achieving complete response (CR), partial response (PR) and stable disease (SD) per RECIST version 1.1. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Week 16
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) Following Single and Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-t) following single (Day 1) and repeat dose (Day 15) administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. The analysis was performed on Pharmacokinetic Population which included all participants in the All Treated Population for whom a pharmacokinetic sample was obtained and analyzed. NA represents data was not available. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Hour*Nanogram per milliliter
  Day 1; n=1, 1, 5, 3, 7, 3, 2, 5, 2 | 10.4 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 21.6 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 32.4 (15.7) | 60.8 (13.8) | 86.0 (57.6) | 190.0 (29.6) | 148.0 (29.9) | 155.2 (29.0) | 129.1 (26.2)
  Day 15; n=1, 1, 5, 1, 5, 3,2, 5,0: number analyzed (Participants) | 1 | 1 | 5 | 1 | 5 | 3 | 2 | 5 | 0
  Day 15; n=1, 1, 5, 1, 5, 3,2, 5,0 | 27.0 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 40.7 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 53.6 (31.5) | 91.1 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 144.1 (64.6) | 122.1 (30.4) | 164.1 (7.8) | 184.4 (40.4) |

12. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) Following Single Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-infinity) following single (Day 1) dose administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 1
Hour*Nanogram per milliliter | 14.5 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 27.2 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 40.0 (18.7) | 70.7 (15.0) | 108.6 (56.1) | 206.3 (27.7) | 163.6 (25.3) | 182.9 (27.1) | 180.9 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation.

13. Secondary Outcome: Part 1: Area Under the Concentration-time Curve Over the Dosing Interval (AUC [0-tau]) Following Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including AUC (0-tau) following repeat (Day 15) dose administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Day 15
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram per milliliter
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 1 | 5 | 3 | 2 | 4 | 0
Hour*Nanogram per milliliter | 27.3 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 40.3 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 53.3 (31.2) | 91.1 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 143.8 (64.2) | 141.9 (32.4) | 164.7 (8.2) | 203.4 (37.2) |

14. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) Following Single and Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including Cmax following single (Day 1) and repeat dose (Day 15) administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Nanogram per milliliter
  Day 1; n=1, 1, 5, 3, 7, 3, 2, 5, 2 | 3.8 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 2.9 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 6.4 (17.3) | 9.3 (12.2) | 12.9 (36.6) | 22.0 (42.9) | 31.2 (26.8) | 23.9 (20.8) | 23.4 (68.8)
  Day 15; n=1, 1, 5, 1, 5, 3, 2, 5, 0: number analyzed (Participants) | 1 | 1 | 5 | 1 | 5 | 3 | 2 | 5 | 0
  Day 15; n=1, 1, 5, 1, 5, 3, 2, 5, 0 | 3.4 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 4.3 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 6.9 (29.2) | 13.8 (NA) — NA indicates the data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 15.7 (39.4) | 15.2 (23.1) | 24.4 (21.5) | 28.1 (7.7) |

15. Secondary Outcome: Part 1: Time to Reach Cmax (Tmax) Following Single and Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including Tmax following single (Day 1) and repeat dose (Day 15) administration of GSK2879552. Tmax is the time to reach Cmax, determined directly from the concentration-time data. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Hours
  Day 1; n=1, 1, 5, 3, 7, 3, 2, 5, 2 | 0.5 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 1.5 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 0.5 (2.8) | 1.3 (110.4) | 0.8 (108.5) | 1.6 (42.5) | 0.8 (85.8) | 1.2 (52.6) | 0.7 (52.1)
  Day 15; n=1, 1, 5, 1, 5, 3, 2, 5, 0: number analyzed (Participants) | 1 | 1 | 5 | 1 | 5 | 3 | 2 | 5 | 0
  Day 15; n=1, 1, 5, 1, 5, 3, 2, 5, 0 | 1.0 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 1.5 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 0.9 (65.1) | 0.5 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 1.1 (88.6) | 1.5 (86.3) | 1.4 (52.1) | 1.0 (46.7) |

16. Secondary Outcome: Part 1: Apparent Terminal Phase Elimination Rate Constant (Lambda z) Following Single and Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including lambda z following single (Day 1) and repeat dose (Day 15) administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available. The data for Day 15 was not computed due to the long half-life of GSK2879552 . Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours^-1
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Hours^-1
  Day 1; n= 1, 1, 5, 3, 6, 3, 2, 5, 1: number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 1
  Day 1; n= 1, 1, 5, 3, 6, 3, 2, 5, 1 | 0.0 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 0.0 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 0.0 (62.6) | 0.1 (8.7) | 0.0 (8.7) | 0.0 (19.1) | 0.1 (47.9) | 0.1 (23.2) | 0.1 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation.
  Day 15; n=0,0,0,0, 0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (T1/2) Following Single and Repeat Dose Administration of GSK2879552
Description: Blood samples were collected from participants for pharmacokinetic analysis including T1/2 following single (Day 1) and repeat dose (Day 15) administration of GSK2879552. Pharmacokinetic analysis of GSK2879552 in Part 1 was conducted by non-compartmental methods. NA represents data was not available. The data for Day 15 was not computed due to the long half-life of GSK2879552. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Hours
  Day 1; n=1, 1, 5, 3, 6, 3, 2, 5, 1: number analyzed (Participants) | 1 | 1 | 5 | 3 | 6 | 3 | 2 | 5 | 1
  Day 1; n=1, 1, 5, 3, 6, 3, 2, 5, 1 | 16.9 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 24.0 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation. | 17.3 (62.6) | 8.8 (8.7) | 18.1 (8.7) | 15.4 (19.1) | 11.5 (47.9) | 8.9 (23.2) | 8.4 (NA) — NA indicates that data was not available since number of participants were insufficient to determine the value for Geometric coefficient of variation.
  Day 15; n=0,0,0,0, 0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Part 1: Accumulation Ratio Following Administration of GSK2879552
Description: The accumulation ratio was analyzed using analysis of variance (ANOVA) for AUC (0-tau) on Day 15 versus AUC (0-tau) on Day 1 by dose cohort. Only dose cohorts with repeat daily dosing were analyzed. The observed accumulation ratio (Ro) was determined based on AUC data to estimate the extent of accumulation after repeat dosing. The Ro of GSK2879552 was estimated by calculating the ratio of the geometric least squares (GLS) means of the pharmacokinetic parameter between Day 15 and Day 1 for all dose levels and the corresponding 90 percent confidence interval (CI) for each ratio.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio of AUC
Arm/Group | Part 1:GSK2879552 1.0 mg Daily | Part 1: GSK2879552 2.0 mg Daily
Number analyzed (Participants) | 5 | 4
Ratio of AUC | 1.917 [1.426 to 2.578] | 1.652 [1.484 to 1.840]

19. Secondary Outcome: Part 1: Time Invariance Ratio Following Administration of GSK2879552
Description: Time invariance was assessed to evaluate whether the pharmacokinetics remains unaltered after repeat dosing. The mixed effect model was fitted with day as a fixed effect and participant as a random effect for each treatment (dose) separately. AUC (0-tau) on Day 15 was compared to AUC (0-infinity) on Day 1 in order to assess time invariance for each dose. The ratio and 90 percent CI were calculated by back-transforming the difference between the LS means for the two days and associated 90 percent CI, for each dose. Only dose cohorts with repeat daily dosing were analyzed.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and Day 15
Population: Pharmacokinetic Population. Only those participants with data available at specific time point were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio of AUC
Arm/Group | Part 1:GSK2879552 1.0 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily
Number analyzed (Participants) | 5 | 5 | 3
Ratio of AUC | 1.332 [1.112 to 1.596] | 1.206 [1.027 to 1.417] | 0.688 [0.412 to 1.149]

20. Secondary Outcome: Part 1: Number of Participants Achieving Disease Control Rate at Week 16
Description: The clinical activity of GSK2879552 given orally in participants with SCLC was evaluated by assessing disease control rate. Clinical response was assessed by the investigator using computer tomography or magnetic resonance imaging scans. Clinical response was defined as disease control rate (CR+PR+SD) based on RECIST version 1.1 at Week 16. Disease control rate was defined as number of participants achieving CR, PR and SD per RECIST version 1.1. The number of participants achieving disease control rate have been presented.
Time Frame: Week 16
Population: All Treated Population.
Measure: Number; unit: Participants
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 7 | 3 | 2 | 5 | 2
Participants | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0

21. Secondary Outcome: Part 1 :Median Effective Dose (ED50) of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and Dose
Description: The pharmacokinetic/pharmacodynamic relationship of GSK2879552 administered orally was characterized by linear and/or non-linear mixed effect models. Only dose cohorts with repeat daily dosing were included in the analysis of platelet as a pharmacodynamic effect. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Percentage change from Baseline was defined as post-dose visit value minus Baseline value, divided by Baseline value and multiplied by 100. Estimates and standard error have been presented.
Time Frame: Baseline and median of 7.286 weeks of drug exposure
Population: Pharmacokinetic Population
Measure: Mean (Standard Error); unit: Milligrams
Groups:
- Part 1: Participants With Repeat Daily Dosing: Participants received repeat daily dosing with GSK2879552 with a starting dose of 0.25 mg once daily for 28 days. The doses were escalated to receive either 0.25 mg or 0.5 or 1 mg or 1.5 or 2 mg or 3 mg daily for 28 days.
Arm/Group | Part 1: Participants With Repeat Daily Dosing
Number analyzed (Participants) | 29
Milligrams | 1.7444 (0.1436)

22. Secondary Outcome: Part 1: ED50 of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and Cmax
Description: The pharmacokinetic/pharmacodynamic relationship of GSK2879552 administered orally was characterized by linear and/or non-linear mixed effect models. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Percentage change from Baseline was defined as post-dose visit value minus Baseline value, divided by Baseline value and multiplied by 100. Only dose cohorts with repeat daily dosing were included in the analysis of platelet as a pharmacodynamic effect. Estimates and standard error have been presented.
Time Frame: Baseline and median of 7.286 weeks of drug exposure
Population: Pharmacokinetic Population
Measure: Mean (Standard Error); unit: Nanogram per milliliter
Arm/Group | Part 1: Participants With Repeat Daily Dosing
Number analyzed (Participants) | 29
Nanogram per milliliter | 10.3948 (1.2666)

23. Secondary Outcome: Part 1: ED50 of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and AUC (0 to Infinity)
Description: as for outcome 22
Time Frame: Baseline and median of 7.286 weeks of drug exposure
Population: Pharmacokinetic Population
Measure: Mean (Standard Error); unit: Hour*Nanogram per milliliter
Arm/Group | Part 1: Participants With Repeat Daily Dosing
Number analyzed (Participants) | 29
Hour*Nanogram per milliliter | 81.8512 (6.0391)

24. Secondary Outcome: Part 2: Number of Participants With SAEs and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Part 2: Number of Participants With DLTs
Description: An event was considered a DLT if it occured within the first 28 days of treatment, and meets one of the following criteria unless it can be clearly established that the event is unrelated to treatment: recurrent Grade 3 anemia after initial transfusion or Grade 3 anemia lasting > 7 days in participants who are not transfused, Grade 4 neutropenia, Grade 3 neutropenia > 7 days duration, febrile neutropenia as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, Grade 3 thrombocytopenia requiring dose reduction, Grade 4 thrombocytopenia lasting > 3 days or of any duration if associated with clinically significant bleeding, drug related Grade 3 or 4 non-hematologic toxicity, drug related Grade 2 toxicity (at any time during treatment) and treatment delay of 14 days or greater due to unresolved drug-related toxicity. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Part 2: Number of Participants With Dose Reduction or Delays
Description: The number of participants who had any dose reduction or delay were planned to be analyzed. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Part 2: Number of Participants Withdrawn Due to Toxicities
Description: Participants were planned to be monitored from start of the study till the development of toxicity in Part 2. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Part 2: Number of Participants With Change in Clinical Chemistry Toxicity Grade From Baseline
Description: Blood samples were planned to be collected for evaluation of clinical chemistry parameters including potassium, aspartate aminotransferase (AST), total bilirubin, creatinine, ALT, uric acid, glucose, GGT, albumin, sodium, calcium, alkaline phosphatase, and phosphorus inorganic. Baseline value was defined as the most recent, non-missing value from a central laboratory prior to or on the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Part 2: Number of Participants With Change in Hematology Toxicity Grade From Baseline
Description: Blood samples were planned to be collected for the analysis of hematology parameters including hemoglobin, lymphocytes, total neutrophils, platelet count and white blood cell (WBC) count. Baseline value was defined as the most recent, non-missing value from a central laboratory prior to or on the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Part 2:Number of Participants With Critical Changes in Values of Vital Signs in Response to Drug
Description: Vital sign measurement includes SBP, DBP, temperature, respiration rate and heart rate. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Part 2: Number of Participants With Abnormal Findings for ECG Parameters
Description: Single measurements of 12-lead ECGs were planned to be obtained in a semi-recumbent or supine position after at least a 5 minutes rest using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Part 2: Number of Participants With Abnormal Findings Undergoing Physical Examinations
Description: The complete physical examination includes assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. A brief physical examination includes assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Part 2: Clearance Following Administration of GSK2879552
Description: Blood samples were planned to be collected for population pharmacokinetic analysis of GSK2879552 including clearance. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Pre-dose, 0.5, and 3 hours post-dose on Day 1; Pre-dose on Day 8; Pre-dose, 0.5 to 1 hour, and 4 to 6 hours on Day 15; Pre-dose at Day 22 and up to every 4 weeks until Week 48
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Part 2: Volume of Distribution Following Administration of GSK2879552
Description: Blood samples were planned to be collected for population pharmacokinetic analysis of GSK2879552 including volume of distribution. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: as for outcome 33
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Part 2: ED50 of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and Dose
Description: The pharmacokinetic/pharmacodynamic relationship of GSK2879552 administered orally was planned to be characterized by linear and/or non-linear mixed effect models. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Percentage change from Baseline was defined as post-dose visit value minus Baseline value, divided by Baseline value and multiplied by 100. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Baseline and up to 2 years
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Groups:
- Part 2 :Participants With Repeat Daily Dosing: Participants with repeat daily dosing were planned to receive GSK2879552 with a starting dose of 0.25 mg once daily for 28 days. The doses were planned to escalate to receive either 0.25 mg or 0.5 or 1 mg or 1.5 or 2 mg or 3 mg daily for 28 days.
Arm/Group | Part 2 :Participants With Repeat Daily Dosing
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 2: ED50 of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and Cmax
Description: as for outcome 35
Time Frame: Baseline and up to 2 years
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2 :Participants With Repeat Daily Dosing
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 2: ED50 of GSK2879552 With Respect to Platelet Nadir as Percent Change From Baseline and AUC (0 to Infinity)
Description: as for outcome 35
Time Frame: Baseline and Up to 2 years
Population: Pharmacokinetic Population. Data was not collected in Part2 as no participant was enrolled in Part2.
Arm/Group | Part 2 :Participants With Repeat Daily Dosing
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 2: Duration of Response
Description: Duration of response for participants is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression or death due to any cause. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of disease progression or death due to any cause. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Part 2: Percentage of Participants Achieving CR and PR
Description: Overall response rate is defined as percentage of participants achieving CR and PR per RECIST version 1.1. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 2 years
Population: All Treated Population. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected in Part 1 from the start of the study treatment up to median of 7.286 weeks of drug exposure.
Description: SAEs and non-SAEs were collected in Part 1 from All Treated Population which included all participants who received at least one dose of study treatment. Data were not collected in Part 2 as no participant was enrolled in Part 2.
Arm/Group | Part 1:GSK2879552 0.25 mg Daily | Part 1:GSK2879552 0.5 mg Daily | Part 1:GSK2879552 1.0 mg Daily | Part 1:GSK2879552 1.5 mg Daily | Part 1: GSK2879552 2.0 mg Daily | Part 1: GSK2879552 3.0 mg Daily | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off | Part 2:GSK2879552 0.25 mg Daily | Part 2:GSK2879552 0.5 mg Daily | Part 2:GSK2879552 1.0 mg Daily | Part 2:GSK2879552 1.5 mg Daily | Part 2: GSK2879552 2.0 mg Daily | Part 2: GSK2879552 3.0 mg Daily | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/5 | 0/3 | 1/7 | 0/3 | 0/2 | 0/5 | 1/2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/5 | 2/3 | 2/7 | 1/3 | 0/2 | 2/5 | 2/2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 5/5 | 2/3 | 6/7 | 3/3 | 2/2 | 5/5 | 1/2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK2879552 0.25 mg Daily (N=1) | Part 1:GSK2879552 0.5 mg Daily (N=1) | Part 1:GSK2879552 1.0 mg Daily (N=5) | Part 1:GSK2879552 1.5 mg Daily (N=3) | Part 1: GSK2879552 2.0 mg Daily (N=7) | Part 1: GSK2879552 3.0 mg Daily (N=3) | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off (N=2) | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off (N=5) | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off (N=2) | Part 2:GSK2879552 0.25 mg Daily (N=0) | Part 2:GSK2879552 0.5 mg Daily (N=0) | Part 2:GSK2879552 1.0 mg Daily (N=0) | Part 2:GSK2879552 1.5 mg Daily (N=0) | Part 2: GSK2879552 2.0 mg Daily (N=0) | Part 2: GSK2879552 3.0 mg Daily (N=0) | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off (N=0) | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off (N=0) | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off (N=0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK2879552 0.25 mg Daily (N=1) | Part 1:GSK2879552 0.5 mg Daily (N=1) | Part 1:GSK2879552 1.0 mg Daily (N=5) | Part 1:GSK2879552 1.5 mg Daily (N=3) | Part 1: GSK2879552 2.0 mg Daily (N=7) | Part 1: GSK2879552 3.0 mg Daily (N=3) | Part 1: GSK2879552 3.0 mg 4 Days on/3 Days Off (N=2) | Part 1: GSK2879552 3.0 mg 4 Days on/10 Days Off (N=5) | Part 1: GSK2879552 4.0 mg 4 Days on/10 Days Off (N=2) | Part 2:GSK2879552 0.25 mg Daily (N=0) | Part 2:GSK2879552 0.5 mg Daily (N=0) | Part 2:GSK2879552 1.0 mg Daily (N=0) | Part 2:GSK2879552 1.5 mg Daily (N=0) | Part 2: GSK2879552 2.0 mg Daily (N=0) | Part 2: GSK2879552 3.0 mg Daily (N=0) | Part 2: GSK2879552 3.0 mg 4 Days on/3 Days Off (N=0) | Part 2: GSK2879552 3.0 mg 4 Days on/10 Days Off (N=0) | Part 2: GSK2879552 4.0 mg 4 Days on/10 Days Off (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (8) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT02034123/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02034123/SAP_001.pdf